CLINICAL TRIAL: NCT01415271
Title: Assessment of an Internet Blood Glucose Management Program in a Chronic Care Hospital
Brief Title: 3-Month Trial Observation of A1c Change
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary exploration of research concept did not prove to be viable.
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, Dr. Hugh Tildesley, Director, Endocrine Research Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Point Grey Trial
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; A1c; internet; long term care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet Intervention (Experimental)
  Interventions: Other: Internet Communication

INTERVENTIONS:
Other: Internet Communication — bi-weekly communication of blood sugars using an internet platform between patients with type 2 diabetes and an endocrinologist

SUMMARY:
The incidence of type 2 diabetes in long term care facilities has been approximated at 25% with barriers to treatment including untimely access to a specialist and improper/poor adherence to insulin regimes. This 3 month trial will investigate the efficacy of improving overall glycemic control by using an internet blood glucose reporting system to facilitate bi-weekly consultations between long term care facility patients with type 2 diabetes and an endocrinologist.

DETAILED DESCRIPTION:
Purpose: This project will investigate the benefits (as measured by change in the primary outcome measure hemoglobin A1c) of bi-weekly reporting of blood sugar values for patients with type 2 diabetes in long term care facilities.

Hypothesis: Our hypothesis is bi-weekly reporting will result in a reduction in A1c after 3 months.

Justification: Elevated A1c values increase risk of health complications for people with type 2 diabetes.

Objectives: Improved type 2 diabetes management for patients in long term care facilities.

Research Methods: Patients who meet the inclusion / exclusion criteria and are interested in participating in the study will self-identify to the research coordinator. Consent will be done in person with any questions answered. Strips and blood glucose meters will be provided. Blood glucose values and testing frequency will be recorded using the internet reporting system Heath-e-Connect. HbA1c, serum creatinine and demographic data will be collected at 0 and 3 months to determine effect of bi-weekly remote communication of blood glucose with an endocrinologist.

Statistical Analysis: HbAlc values at 0 and 3 months will be compared using an unpaired t-test to measure the effect of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus patients at Point Grey Private Hospital
* Trained in self-blood glucose monitoring
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be trained on IBGMS

Exclusion Criteria:

* Patients with medical conditions that may affect their study participation or results will be excluded.
* Patients currently being treated with steroid medication
* Patients that have impaired liver function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | 0 and 3 months
  Hemoglobin A1c will be measure at 0 and 3 months to determine the efficacy of the internet blood glucose monitoring system as measured by change in glycemic control.

SECONDARY OUTCOMES:
Staff satisfaction | 3 months
  Measure of hospital staff satisfaction of using the Health-e-Connect platform to help patients communicate with an endocrinologist
Frequency of Self-Monitoring | 3 months
  Measure the frequency of blood glucose self-monitoring of the patients by collecting the total number of tests using the provided meter.
unplanned hospitalizations | 3 months
  A secondary endpoint includes adverse events such as unplanned hospitalizations for any cause that last more than 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Tildesley, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- Endocrine Research Society, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Clement M and Leung F. Diabetes and the Frail Elderly in Long-term Care. Can J Diabetes. 2009;33(2):114-121.
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] American Diabetes Association. Standards of medical care in diabetes--2008. Diabetes Care. 2008 Jan;31 Suppl 1:S12-54. doi: 10.2337/dc08-S012. No abstract available. PMID 18165335
- [Background] Karter AJ, Ackerson LM, Darbinian JA, D'Agostino RB Jr, Ferrara A, Liu J, Selby JV. Self-monitoring of blood glucose levels and glycemic control: the Northern California Kaiser Permanente Diabetes registry. Am J Med. 2001 Jul;111(1):1-9. doi: 10.1016/s0002-9343(01)00742-2. PMID 11448654
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Tildesley HD, Mazanderani, AB, Chan, JHM et al. Efficacy of A1c Reduction Using Internet Intervention in Patients with Type 2 Diabetes Treated with Insulin. Can J Diabetes. 2011; 35(3): 250-253.